CLINICAL TRIAL: NCT00462410
Title: Socio-anthropological Study Evaluating the Impact of Observance or Treatment in Patients With Breast Cancer
Brief Title: Effect of Advertisements on Treatment Compliance in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Health Services Research
Other Study IDs: CDR0000540528; IB-2006-03; INCA-REF0145; INCA-SOCIO-ANTHROPO
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Psychiatric Rehabilitation

INTERVENTIONS:
Other: counseling intervention
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Measuring how advertising affects treatment compliance in women with breast cancer may help doctors plan the best treatment.

PURPOSE: This clinical trial is studying how advertisements affect treatment compliance in women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the consequences of advertisement on treatment compliance in women with breast cancer.

Secondary

* Determine the factors favoring or not favoring adherence to the medical recommendations.

OUTLINE: Patients and their medical and nonmedical caregivers are interviewed by a sociologist or anthropologist twice over 1 year. The first interview is at the consultation visit and the second interview is at the patient's home. The impact of advertisement on treatment compliance is measured.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Treatment compliance

SECONDARY OUTCOMES:
Factors affecting adherence to the medical plan

CONTACTS AND LOCATIONS:
Overall Officials: Marc Debled, MD, Study Chair — Institut Bergonié